CLINICAL TRIAL: NCT02572934
Title: Health Status and Burden of Late Effects in Very Long-term Testicular Cancer Survivors (STANDBY-study)
Acronym: STANDBY
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL53126.042.15
Record Dates: First submitted 2015-08-27; First posted 2015-10-09 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Testicular Cancer
Keywords: Testicular cancer; Survivorship; late adverse treatment effects
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Chemotherapy group (CT-group): Patients treated with chemotherapy >20 years ago
- Radiotherapy group (RT-group): Patients treated with radiotherapy >20 years ago
- Surgery-only group (SU-group): Patients treated with only orchidectomy >20 years ago
- Control-group: Healthy controls

SUMMARY:
Depending on disease stage, testicular cancer (TC) treatment consists of an orchidectomy, alone or followed by radiotherapy (RT) or platinum-based chemotherapy (CT). TC survival rates are above 90% nowadays, which results in growing TC survivor population. Because of the long life expectancy of these survivors, prevention or early detection of late treatment effects has become increasingly relevant. Yet known late effects are nephrotoxicity, cardiovascular disease (CVD), secondary malignant neoplasms (SMN), neurotoxicity, pulmonary toxicity, Raynaud's phenomenon, hypogonadism, fatigue and psychosocial problems. Nephrotoxicity is an important late effect, but data is lacking in very long-term survivors since performed studies have a follow-up duration of 5-14 years. Decreased renal function is a known risk factor for CVD development and also an association between renal function and neurtoxicity via circulating platinum levels has been shown. It is hypothesized that treatment induced nephrotoxicity is prevalent in TC survivors and might be a mediator for development of late effects. The secondary aim is to assess prevalence of late effects in very long-term TC survivors: until now, most data have been collected through questionnaires in large epidemiological studies in TC survivors till approximately 10 years after treatment. The prevalence of late effects may increase over time: 10 years after treatment late effects may not be present yet, whilst late effects can emerge just after 20 years. Consequently, health status and possible late effects, resulting in morbidity, are underestimated in patients who are 20-30 years after treatment. By investigating health status of these very long-term survivors a more profound insight in the prevalence and aetiology of these late effects and the development over time can be assessed. Current treatment is very similar to TC treatment 20-30 years ago and therefore knowledge on late effects is relevant for currently treated patients. Furthermore, as a result of this study, we will better understand which factors and issues should be watched closely during follow-up, which TC survivors are at increased risk of developing late treatment effects and how to detect early damage before overt morbidity occurs.

DETAILED DESCRIPTION:
Objective: The aim of this study is to compare glomerular filtration rate (GFR) in very long-term testicular cancer (TC)-survivors treated with chemotherapy, radiotherapy or surgery only and non-cancer treated healthy controls. Secondary aim is to assess prevalence of adverse late treatment effects in very long-term TC-survivors treated with chemotherapy (CT), radiotherapy (RT) or surgery only (SU) and investigate the relationship between GFR parameters and these late effects.

Study population: Patients treated with CT, RT or only surgery for TC more than 20 years ago and an age-matched male control population.

Study design: An observational cross-sectional cohort study will be performed. Patients will be invited for a single study visit, which consists of collection of urine during 24 hours, withdrawal of blood samples, filling in questionnaires, physical examination, vascular function and structure tests, lung function tests, digital cooling tests, neuropsychological assessment and a walk test.

Main study parameters/endpoints: Primary study parameter is renal function as expressed by glomerular filtration rate (GFR). Secondary endpoints are the prevalence of the following defined adverse late effects: cardiovascular disease (CVD), peripheral neuropathy, reduced lung function, Raynaud's phenomenon, hypogonadism, fatigue and cognitive dysfunction. Other secondary parameters are health related quality of life (HRQoL), physical fitness, markers for (subclinical) vascular damage, single nucleotide polymorphisms (SNPs) and aging markers.

ELIGIBILITY:
Inclusion Criteria:

1. Age <70 years at time of inclusion
2. Signed informed consent
3. CT-, RT- and SU-group: Age at start of TC treatment <40 yrs.
4. CT-, RT- and SU-group: At least 20 years after start of treatment for TC at time of inclusion.
5. CT-group: Patients treated with cisplatin-based chemotherapy for TC with good or intermediate prognosis (according to IGCCCG prognosis group).
6. RT-group: Patients treated with radiotherapy for TC stage I or II.
7. SU-group: Patients treated with orchidectomy only for TC stage I.

Exclusion Criteria:

1. Mental disorder (no informed consent available).
2. CT-group: Patients also treated with radiotherapy for TC.
3. RT-group: Patients also treated with chemotherapy for TC.
4. SU-group: Patients also treated with chemo- or radiotherapy for TC.
5. CO-group: Treated with chemotherapy, radiotherapy or hormonal therapy for any type of cancer.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participating TC survivors will be identified by the TC registry of the uro-oncology tumor working group of the UMCG. The investigators will randomly select (with an SPSS-query) 70 potential participants from the CT-group and search for age-matched controls in the RT-, SU- and CO-group. A margin of three years will be accepted. If no matching RT-patients, SU-patients or healthy volunteers are available, age-matching criteria will be relaxed by allowing the difference to increase with one year at each step, to a maximum of six years. Vital status will be checked with help of information from the municipal population registry (GBA:'gemeentelijke basisadministratie'). Healthy volunteers are recruited via advertisements in local door-to-door papers and by flyers exposed in the UMCG.
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) in ml/min | 3 years

SECONDARY OUTCOMES:
Development of cardiovascular disease (CVD) according to the WHO ICD-10 classification (I10-I15: hypertensive disease; I20-I25: ischemic heart disease; I60-I69: cerebrovascular disease; I70-I79: disease of arteries, arterioles and capillaries) | 3 years
Peripheral neuropathy (anamnestic with SCIN questionnaire which assesses a.o. chemotherapy-induced peripheral sensory neuropathy) | 3 years
Raynaud's phenomenon (anamnestic with SCIN questionnaire which assesses a.o. Raynaud's phenomenon and objectified with standardized digital cooling tests) | 3 years
Lung function (FEV1, FVC, TLC, RV, FRC and diffusion capacity (DLCO, KCO)) | 3 years
Hypogonadism (LH > 10 U/l or testosterone < 14 ng/ml) | 3 years
Cognitive function (neuropsychological assessment of different domains: learning, memory, processing speed, executive function) | 3 years
Fatigue (scaled; VVV-questionnaire) | 3 years
Testicular cancer disease characteristics: stage, prognosis group, chemotherapy regimen/dose, radiotherapy doses/location | 3 years
Health-related quality of life (HRQoL) | 3 years
Physical fitness (according to six-minute walk test with sex, age and BMI specific reference values) | 3 years
Intima media thickness (IMT) | 3 years
Advanced Glycation End products (AGEs) | 3 years
Cardiovascular risk factors (presence of hypertension, dyslipidemia, impaired fasting glucose, overweight/obesity, tobacco and alcohol use, family history) | 3 years
Genetic susceptibility for (cardio)vascular damage (single nucleotide polymorphisms (SNPs) in DNA) | 3 years
Leukocyte telomere length | 3 years
Arterial stiffness measured as pulse-wave velocity (PWV) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jourik Gietema, MD PhD, Principal Investigator — Universirty Medical Centre Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stelwagen J, Meuleman AT, Lubberts S, Steursma G, Kruyt LM, Donkerbroek JW, Meijer C, Walenkamp AME, Lefrandt JD, Rakers SE, Huitema RB, de Jong MAA, Wiegman EM, van den Bergh ACM, de Jong IJ, van Rentergem JAA, Schagen SB, Nuver J, Gietema JA. Cognitive Impairment in Long-Term Survivors of Testicular Cancer More Than 20 Years after Treatment. Cancers (Basel). 2021 Nov 12;13(22):5675. doi: 10.3390/cancers13225675. PMID 34830829
- [Derived] Stelwagen J, Lubberts S, Steggink LC, Steursma G, Kruyt LM, Donkerbroek JW, van Roon AM, van Gessel AI, van de Zande SC, Meijer C, Grafin Zu Eulenburg CH, Oosting SF, Nuver J, Walenkamp AME, Jan de Jong I, Lefrandt JD, Gietema JA. Vascular aging in long-term survivors of testicular cancer more than 20 years after treatment with cisplatin-based chemotherapy. Br J Cancer. 2020 Nov;123(11):1599-1607. doi: 10.1038/s41416-020-01049-3. Epub 2020 Sep 14. PMID 32921790